CLINICAL TRIAL: NCT07318896
Title: Evaluation of the Effect of Agar and/or Collagen Based Compounds on Osteoarticular Pain. A Randomized, Parallel, Placebo Controlled, Triple Blind Clinical Trial (AGARTROSIS)
Brief Title: Effect of Agar/Collagen-based Compounds on Osteoarticular Pain: Randomized Triple-blind Clinical Trial
Acronym: AGARTROSIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: HISPANAGAR SA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGARTROSIS
Record Dates: First submitted 2025-11-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Osteearthritis; Joint Damage; Inflammation; Cartilage Damage
Keywords: Agar-Agar; undenatured collagen type II; Joint pain; knee pain
MeSH Terms: conditions — Inflammation; Arthralgia | interventions — Agar

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, placebo-controlled, triple-blind nutritional intervention clinical study, with a 1:1:1:1 ratio between interventions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Agar-Agar (A-A) (Experimental): Participants assigned to this group will receive agar-agar (A-A) supplementation and will take it for 12 weeks.
  Interventions: Dietary Supplement: Agar-Agar
- Agar-Agar + undenatured collagen type II (A+UC-II) (Experimental): Participants assigned to this group will receive agar-agar and undenatured collagen type II (A+UC-II) supplementation and will take it for 12 weeks.
  Interventions: Dietary Supplement: Agar-Agar and undenatured collagen type II
- undenatured collagen type II (UC-II) (Active Comparator): Participants assigned to this group will receive undenatured collagen type II (UC-II) supplementation and will take it for 12 weeks.
  Interventions: Dietary Supplement: undenatured collagen type II
- Placebo (Placebo Comparator): Participants assigned to this group will receive the placebo and will take it for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Agar-Agar — 2.4 g of agar-agar (Rhodophyceae group) presented in capsule form will be given.
  Other Names: (A-A)
  Arms: Agar-Agar (A-A)
Dietary Supplement: Agar-Agar and undenatured collagen type II — 2.4 g of agar- agar + 40 mg of undenatured collagen type II, presented in capsule form will be given.
  Other Names: (A+UC-II)
  Arms: Agar-Agar + undenatured collagen type II (A+UC-II)
Dietary Supplement: undenatured collagen type II — 40 mg of undenatured collagen type II + 2.4 g of maltodextrin will be given in capsule form
  Other Names: (UC-II)
  Arms: undenatured collagen type II (UC-II)
Dietary Supplement: Placebo — 2.4 g Maltodextrin will be given in capsule form
  Arms: Placebo

SUMMARY:
Joints-comprising bone, cartilage, ligaments, and synovial fluid-enable stable daily movement but may deteriorate with age, excess body weight, overuse, injury, or disease. Such degeneration, common from age 40 onward, underlies joint disorders like osteoarthritis, particularly in the knees, hips, hands, and spine, and is a major cause of chronic pain and disability. While antiinflammatory analgesics remain the standard approach to symptom control, they neither cure disease nor regenerate cartilage and can produce significant long-term adverse effects (gastrointestinal, hepatic, renal, and cardiovascular). These limitations motivate interest in natural or complementary strategies with safer profiles.

Within this context, marine algae, especially agar derived from red seaweed, have attracted attention for potential intestinal, metabolic, and joint benefits, aided by their fiber content. Another promising option is undenatured type II collagen (UC-II), the principal structural component of articular cartilage, whose endogenous production declines with age; clinical studies indicate that a daily intake of 40 mg UC-II can improve mobility, reduce pain, and enhance quality of life in individuals with osteoarthritis or exercise-related joint discomfort. Based on these considerations, an agar-agar supplement has been developed to relieve knee joint symptoms.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the effect of agar-agar (A-A), the combination of A-A with undenatured type II collagen (A+UC-II), and undenatured type II collagen (UC-II) on knee joint pain, assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), in subjects with mild to moderate joint pain without a diagnosis of osteoarthritis, compared with a control compound.

The secondary objectives were to evaluate the effects of A-A, A+UC-II, and UC-II consumption on:

* Knee joint stiffness and functional capacity (subjective assessment).
* Overall perception of knee health (subjective assessment).
* Pain, stiffness, and functional capacity of the hand (subjective assessment).
* Range of motion of the knee.
* Functional capacity of the knee (objective assessment).
* Functional capacity of the hand (objective assessment).
* Frequency of medication use for joint pain relief (anti-inflammatories, analgesics).
* Inflammatory blood markers.
* Blood markers of collagen and bone metabolism.
* Body composition.

The primary endpoint is patient-reported knee joint pain, assessed using the Pain subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire.

This is a randomized, placebo-controlled, triple-blind, parallel-group nutritional intervention with an allocation ratio of 1:1:1:1. A total of 80 participants (men and women) will be enrolled. Following a pre-screening visit to verify inclusion and exclusion criteria, eligible participants will be randomly assigned to one of four groups (n=20 per group) to consume, once daily for 12 weeks, one of the following products: agar-agar (A-A), A-A+UC-II (A+UC-II), UC-II alone, or placebo.

Each participant will complete three in-person visits and one interim telephone follow-up: a pre-screening visit (eligibility assessment), a baseline visit to initiate the intervention, a mid-study telephone follow-up, and an end-of-study visit. The total duration per participant will be 13 weeks.

The primary endpoint is patient-reported knee joint pain, assessed using the Pain subscale of the WOMAC questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 40 and 70 years of age.
* Submit a score of 6 to 10 out of 20 on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) knee pain questionnaire.
* Sign the informed consent form.
* Know how to read, write, and speak Spanish and/or Catalan.

Exclusion Criteria:

* Present body mass index (BMI) values <18.5 kg/m^2 or ≥30 kg/m^2.
* Present intolerances or allergies related to Agar-Agar, or any of the components of the products being evaluated, such as collagen or maltodextrin.
* Take or have taken medications that may affect the study results. This is especially true for those who have been treated with oral or intra-articular corticosteroids within the 4 and 12 weeks prior to screening, respectively, or medications for osteoarthritis at the time of screening.
* Patients who depend on prescription medications for pain control.
* Take multivitamin or mineral supplements, collagen derivatives, or supplements containing bioactive compounds that may exert an anti-inflammatory effect, such as turmeric, ginger, omega-3, or polyphenol supplements.

(Individuals who consume multivitamin, mineral, or collagen-derived supplements or supplements will be eligible to participate in the study, provided they are willing to discontinue their intake for at least two weeks prior to the start of the study and throughout the entire study period).

* Be an active smoker or have been one for less than 6 months.
* Alcohol consumption:

  * Men: Consume 4 or more Standard Drink Units (SDU) daily or SDUs weekly.
  * Women: Consume 2 or more Standard Drink Units (SDU)* daily or SDUs weekly.
* Have a diagnosis of osteoarthritis, active rheumatoid arthritis, and any inflammatory arthritic condition such as secondary inflammatory arthritis, gout, pseudogout, knee infection, marked angular deformities, or significant injury to the target joint within the 6 months prior to the start of the trial; arthroplasty and joint surgery of the target knee within the 2 years prior to the start of the study.
* Have any gastrointestinal disease that affects the absorption of the compound and/or the study results, such as celiac disease, Crohn's disease, active cancer of any organ of the digestive or renal system, or hepatitis.
* Be ineligible to participate in the study, according to the pre-screening evaluator's criteria.
* Have lost 3 kg or more in the last 3 months.
* Be pregnant or intend to become pregnant.
* Be breastfeeding.
* Be unable to follow the study guidelines.
* Be participating or have participated in a clinical trial involving drug intervention or nutritional intervention within the last 30 days prior to inclusion in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in perception of knee joint pain. | Before (baseline), during (6 weeks) and after treatment period (12 weeks).
  This will be determined using the pain subscale of the Western Ontario and McMaster Universities Osteoarthritis Index questionnaire.
  The questionnaire assesses clinically meaningful changes in symptoms and physical disability in individuals with osteoarthritis or those experiencing joint discomfort. It evaluates the perceived intensity of knee pain using the Likert scale (0: no pain; 1: mild pain; 2: moderate pain; 3: severe pain; 4: extreme pain).

SECONDARY OUTCOMES:
Body weight. | at week 1.
  Body weight will be measured by Tanita TBF-300 (Body Composition Analyzer, Brooklyn NY, USA) as a descriptive variable.
Height. | At week 1.
  Height will be measured by standardized method.
Body mass index (BMI) (kg/m^2). | At week1.
  BMI will be determined using the Tanita TBF-300 (Body Composition Analyzer, Brooklyn, NY, USA) as a descriptive variable.
Age. | At week 1.
  Age will be recorded in years.
Changes in systolic and diastolic blood pressure and resting heart rate. | Before (baseline) and after treatment period (12 weeks).
  It will be measured using an automatic sphygmomanometer.
Changes in body weight. | Before (baseline) and after treatment period (12 weeks).
  Body weight will be measured by Inbody 970.
Change in BMI. | Before (baseline) and after treatment period (12 weeks).
  Weight and height will be combined to report BMI in kg/m^2.
Changes in the amount of body fat. | Before (baseline) and after treatment period (12 weeks).
  Body fat in kg will be measured with Inbody 970.
Changes in the amount of body fat. | Before (baseline) and after treatment period (12 weeks).
  Body fat percentage will be measured with Inbody 970.
Changes in the amount of muscle mass. | Before (baseline) and after treatment period (12 weeks).
  Muscle mass in kg will be measured by Inbody 970.
Changes in the amount of muscle mass. | Before (baseline) and after treatment period (12 weeks).
  Muscle mass percentage will be measured by Inbody 970.
Changes in the amount of bone mass. | Before (baseline) and after treatment period (12 weeks).
  Bone mass (kg) will be measured by Inbody 970.
Changes in the amount of total body water. | Before (baseline) and after treatment period (12 weeks).
  Total body water (Kg) will be measured by Inbody 970.
Change in the amount of lean mass. | Before (baseline) and after treatment period (12 weeks).
  The total lean mass (Kg) will be measured by Inbody 970.
Changes in bone mineral content. | Before (baseline) and after treatment period (12 weeks).
  This will be measured, in Kg, by Inbody 970.
Changes in segmental impedance. | Before (baseline) and after treatment period (12 weeks).
  This will be measured by Inbody 970.
Changes in segmental phase angle. | Before (baseline) and after treatment period (12 weeks).
  The phase angle (kHz) will be measured by Inbody 970.
Change in perception of knee joint stiffness. | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the rigidity subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire. It consists of two items. The perceived intensity of knee stiffness will be evaluated in two different situations: in the morning, immediately after waking up, and during the day, following a period of rest or inactivity, using the Likert scale (0: no stiffness; 1: mild stiffness; 2: moderate stiffness; 3: severe stiffness; 4: extreme stiffness) (total scale 0-8).
Change in perception of knee functional capacity. | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the rigidity subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire.
  It consists of 17 items. The difficulty in performing various activities-such as climbing or descending stairs, walking, bending, or carrying out daily tasks-will be evaluated using the Likert scale (0: no difficulty; 1: mild difficulty; 2: moderate difficulty; 3: severe difficulty; 4: extreme difficulty) (total scale 0-68).
Changes in the perception of the general health status of the knee | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the rigidity subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questionnaire.
  It will be obtained by summing the scores of the three subscales: pain, stiffness, and physical function. The total score ranges from 0 to 96, reflecting the best and worst possible knee condition, respectively.
Perception of pain in the hand joint | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the pain subscale of the Australian-Canadian Hand Osteoarthritis Index (AUSCAN) questionnaire. The questionnaire consists of 5 items that assess, over the previous 48 hours, the intensity of pain at rest and while grasping, lifting, turning, and squeezing objects, using a Likert scale (0: no pain; 1: mild pain; 2: moderate pain; 3: severe pain; 4: extreme pain).
Changes in perception of hand joint stiffness | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the pain subscale of the Australian-Canadian Hand Osteoarthritis Index (AUSCAN) questionnaire. It consists of 1 item that assesses, over the previous 48 hours, the intensity of hand stiffness upon waking, using a Likert scale (0: no stiffness; 1: mild stiffness; 2: moderate stiffness; 3: severe stiffness; 4: extreme stiffness).
Changes in perception of the functional capacity of the hand joint | Before (baseline) during ( 6 weeks) and after treatment period (12 weeks).
  This variable will be assessed using the pain subscale of the Australian-Canadian Hand Osteoarthritis Index (AUSCAN) questionnaire. It consists of 7 items that assess, over the previous 48 hours, the difficulty in turning, holding, opening, carrying, grasping, and squeezing various objects with the hand, using a Likert scale (0: no difficulty; 1: mild difficulty; 2: moderate difficulty; 3: severe difficulty; 4: extreme difficulty).
Changes in knee range of motion | Before (baseline) and after treatment period (12 weeks).
  This variable will be measured using a digital goniometer.
Changes in the functional capacity of the hand joints | Before (baseline), and after treatment period (12 weeks)
  Hand grip strength will be measured, in kilograms, using the InGrip digital dynamometer.
Changes in the speed when going up and down stairs. | Before (baseline) and after treatment period (12 weeks).
  This variable will measured by The "Stair Climb Test" , in which the volunteer must climb and descend 10 standard steps (between 15 and 20 cm) without the aid of a handrail. The time (minutes and seconds) taken by the volunteer to complete the test will be recorded.
Changes in pain perception at the end of the Stair Climb Test | Before (baseline) and after treatment period (12 weeks).
  At the end, perceived pain will be measured using a 100 mm visual analog scale, where 0 indicates "no pain" and 100 indicates "all the pain you can experience".
Changes in plasma interleukin 6 (IL-6) concentration. | Before (baseline) and after treatment period (12 weeks).
  Plasma IL-6 levels will be measured by ELISA kits
Changes in plasma tumor necrosis alpha (TNF-a) concentration. | Before (baseline) and after treatment period (12 weeks).
  Plasma TNF-a levels will be measured by ELISA kit.
Changes in plasma monocyte chemotactic protein 1 (MCP-1) concentration | Before (baseline) and after treatment period (12 weeks).
  Plasma MCP-1 levels will be measured ELISA kit.
Changes in serum High-sensitivity C-reactive protein (hsCRP) concentration. | Before (baseline) and after treatment period (12 weeks).
  Serum hsCRP levels will be measured by chemiluminescence method.
Changes in serum levels of C-terminal telopeptide of type 1 collagen (CTX1). | Before (baseline) and after treatment period (12 weeks).
  Serum CTX1 will be measured by electrochemiluminescence method.
Changes in serum levels of N-terminal propeptide of type I collagen (PINP). | Before (baseline) and after treatment period (12 weeks).
  Serum PINP will be measured by electrochemiluminescence method.
Changes in serum levels of hyaluronic acid (HA). | Before (baseline) and after treatment period (12 weeks).
  Serum HA will be measured by ELISA kits.
Changes in serum levels of cartilage oligomeric matrix protein (COMP). | Before (baseline) and after treatment period (12 weeks).
  Serum COMP will be measured by ELISA kits.
Dietary control. | Before (baseline), during (6 week) and after treatment period (12 weeks).
  The intake of foods containing bioactive components that could alleviate pain will be assessed using an adapted food frequency questionnaire.
  The following scale will be used: "I have not used it"; "1 time a week"; "2-4 times a week"; "5-6 times a week"; "7-10 times a week"; "10-20 times a week"; ">20 times a week"
Changes in dietary supplement use. | Before (baseline), during (6 week) and after treatment period (12 weeks).
  The consumption of supplements and dietary products by the volunteers will be monitored through the analysis of the supplement and dietary product records in the case report form.
Changes in concomitant medications. | Before (baseline), during (6 week) and after treatment period (12 weeks).
  The consumption of concomitant medication will be monitored through the analysis of the concomitant medication records in the case report form.
Changes in pain-relieving medication use. | Before (baseline), during (6 week) and after treatment period (12 weeks).
  This will be assessed by recording concomitant medications in the data collection form.
Physical activity levels. | Before (baseline), and after treatment period (12 weeks).
  This will be determined by analyzing the Physical Activity Questionnaire, Quick Physical Activity Classifier, adapted from the Generality of Catalonia (PEFS) guidelines.
Monitoring of adverse effects. | During (6 week) and after treatment period (12 weeks).
  The presence of adverse events reported by the participant in the data collection form will be recorded using the Adverse Effects Form.
Treatment adherence rate. | During (6 week) and after treatment period (12 weeks).
  Treatment adherence will be calculated using the following formula: (number of capsules the volunteer should have taken / number of capsules actually taken) * 100

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari Palou, PhD, Principal Investigator — UTNS (Eurecat, Reus)
Locations (1):
- Eurecat, Technological Center of Catalonia, Nutrition and Health Unit, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus — http://eurecat.org